CLINICAL TRIAL: NCT03111589
Title: Monocytic Expression of Heme Oxidase-1 (HO-1) in Sickle Cell Patients and Correlation With the Humoral Immune Response to Vaccine and With Allo-immunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francis Corazza (Other)
Responsible Party: Sponsor-Investigator, Francis Corazza, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUB-HO1 sickle cell
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Heme oxidase-1 (HO-1)
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCD patients under regular chronic exchange transfusion (Experimental): Sickle cell disease patients (SCD) under regular chronic exchange transfusions. Pediatric and adult patients from the HUDERF and CHU-Brugmann Hospitals.
  Interventions: Biological: Inactivated influenza A (H1N1) virus vaccine; Diagnostic Test: Blood sampling
- SCD patients under HU treatment alone (Experimental): Sickle cell disease patients (SCD) under hydroxyurea (HU) alone. Pediatric and adult patients from the HUDERF and CHU-Brugmann Hospitals.
  Interventions: Biological: Inactivated influenza A (H1N1) virus vaccine; Diagnostic Test: Blood sampling
- SCD patients under HU treatment+sporadic transfusion (Experimental): Sickle cell disease patients (SCD) under hydroxyurea (HU) and receiving sporadic transfusions.Pediatric and adult patients from the HUDERF and CHU-Brugmann Hospitals.
  Interventions: Biological: Inactivated influenza A (H1N1) virus vaccine; Diagnostic Test: Blood sampling
- Control group (Active Comparator): Pediatric and adult patients from the HUDERF and CHU-Brugmann Hospitals.
  Interventions: Biological: Inactivated influenza A (H1N1) virus vaccine; Diagnostic Test: Blood sampling

INTERVENTIONS:
Biological: Inactivated influenza A (H1N1) virus vaccine — All groups of patients and the control group will receive the new annually recommended inactivated influenza A (H1N1) virus vaccine.
Diagnostic Test: Blood sampling — Testing of the different humoral immune responses to vaccines or to erythrocyte alloantigens.

SUMMARY:
Sickle cell disease (SCD) is an autosomal recessive disorder resulting from a substitution in the β chain of hemoglobin (Hb) which causes hemoglobin S to polymerize when deoxygenated. SCD patients present immune abnormalities that have always been attributed to functional asplenia. It it is now being recognized that patients with SCD have a pro-inflammatory condition with altered immune system activation contributing to the pathology of SCD. Increased levels of neutrophils, monocytes or cytokines have been reported in SCD patients.

SCD is associated with many acute and chronic complications requiring immediate support. Actual strongly recommended therapies include chronic blood transfusions (CT) and hydroxyurea (HU). In addition, episodic transfusions are recommended and commonly used to manage many acute SCD complications.There is strong evidence to support the use of HU in adults with 3 or more severe vaso-occlusive crises during any 12-month period, with SCD pain or chronic anemia, or with severe or recurrent episodes of acute chest syndrome. HU use is now also common in children with SCD. Some patients receive chronic monthly RBC transfusion with the objective to reduce the proportion of HbS to < 30 %. Long-term RBC transfusions prevent and treat complications of SCD decreasing the risk of stroke and the incidence of acute chest syndrome (ACS).

Therapeutic complications, such as alloimmunization against RBC in 20-50% of patients or hematopoietic stem cell transplantation (HSCT) graft rejection, constitute an immune-based clinical issue in SCD. Poorly understood RBC alloimmunization is responsible for serious hemolytic transfusion reaction associated with severe mortality and morbidity underlying the need for a better understanding of the immunology of SCD to improve SCD transfusion support/outcome. Little evidence exists about HU effects on immune functions in SCD. HU treatment doesn't appear to have deleterious effects on immune function and appears to decrease the abnormally elevated number of total WBC and lymphocytes, while CT does not.

Patients with SCD are at higher risk of infections and prophylactic vaccination is strongly recommended. Recent data suggest that vaccinal response to pneumococcal antigens in SCD patients is identical to healthy control while controversy concern the stability of the immune protection after vaccination of SCD patient. Antibody levels declined over the year and the need for more frequent vaccination in SCD patient should be investigated. Currently, there is no evidence whether HU may interfere with pneumococcal immune response. Purohit showed that immune response to inactivated influenza A (H1N1) virus vaccine was altered in patient with SCD receiving CT but little is known on immune response to vaccination in patients with SCD receiving HU.

Recent data suggest that not only inflammatory status but also humoral immune response to antigens in SCD patients may differ according to treatment. Yazdanbakhsh reported an imbalance between regulatory T cell (Treg) and effector T cell (Teff) in alloimmunized SCD patients with as consequence an increase in antibody production. In a model proposed by the authors, the balance between Treg and Teff is dictated by the monocyte control of cytokines expression. Altered activity of monocyte heme oxidase-1 (HO-1) would be responsible of a decrease in IL-12 and an increase in IL-10 cytokines secretion impacting the Treg/Teff cells ratio and promoting antibody production by B cells.

The objectives of the project are to assess whether different humoral immune responses to vaccines or to erythrocyte alloantigens are related to the type of treatment administered to patients with SCD. We also aim to study if these differences might be related to different expressions of HO-1 by monocytes.

ELIGIBILITY:
Inclusion Criteria:

- Pediatric and adult patients with sickle cell disease from the HUDERF and CHU-Brugmann Hospital

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Intracellular HO-1 expression in monocytes | 1 month post vaccination
  Intracellular monocyte heme oxidase-1 (HO-1) expression will be measured by flow cytometry.The protein expression of HO-1 will be confirmed by Western blot. A commercial ELISA kit will be used in parallel to assess HO-1 levels in PBMC cell lysate.
HO-1 level in serum | 1 month post vaccination
  Monocyte heme oxidase-1 (HO-1) level in serum will be measured by a commercial ELISA kit
Cytokines levels measurement | 1 month post vaccination
  Pro-inflammatory cytokine (IL-12) and anti-inflammatory cytokine (IL-10) levels will be evaluated in serum and in IL-1 stimulated whole blood supernatants using an ELISA assay.
Identification of T regulatory cells | 1 month post vaccination
  Evaluation of Treg cells in peripheral blood mononuclear cells (PBMC) will be performed by flow cytometry using appropriate fluorochrome conjugated monoclonal antibodies for CD25 and FoxP3 markers
Immune response to vaccination | 1 month post vaccination
  Post-vaccination serum H1N1 antibodies titers (IgG and IgM) will be measured by an ELISA kit

SECONDARY OUTCOMES:
Intracellular HO-1 expression in monocytes | Baseline: at vaccination
  Intracellular HO-1 expression will be measured by flow cytometry.The protein expression of HO-1 will be confirmed by Western blot. A commercial ELISA kit will be used in parallel to assess HO-1 levels in PBMC cell lysate.
Intracellular HO-1 expression in monocytes | 3 months post vaccination
  Intracellular HO-1 expression will be measured by flow cytometry.The protein expression of HO-1 will be confirmed by Western blot. A commercial ELISA kit will be used in parallel to assess HO-1 levels in PBMC cell lysate.
Intracellular HO-1 expression in monocytes | 6 months post vaccination
  Intracellular HO-1 expression will be measured by flow cytometry.The protein expression of HO-1 will be confirmed by Western blot. A commercial ELISA kit will be used in parallel to assess HO-1 levels in PBMC cell lysate.
HO-1 level in serum | Baseline: at vaccination
  HO-1 level in serum will be measured by a commercial ELISA kit
HO-1 level in serum | 3 months post vaccination
  HO-1 level in serum will be measured by a commercial ELISA kit
HO-1 level in serum | 6 months post vaccination
  HO-1 level in serum will be measured by a commercial ELISA kit
Cytokines levels measurement | Baseline: at vaccination
  Pro-inflammatory cytokine (IL-12) and anti-inflammatory cytokine (IL-10) levels will be evaluated in serum and in IL-1 stimulated whole blood supernatants using an ELISA assay.
Cytokines levels measurement | 3 months post vaccination
  Pro-inflammatory cytokine (IL-12) and anti-inflammatory cytokine (IL-10) levels will be evaluated in serum and in IL-1 stimulated whole blood supernatants using an ELISA assay.
Cytokines levels measurement | 6 months post vaccination
  Pro-inflammatory cytokine (IL-12) and anti-inflammatory cytokine (IL-10) levels will be evaluated in serum and in IL-1 stimulated whole blood supernatants using an ELISA assay.
Identification of T regulatory cells | Baseline: at vaccination
  Evaluation of Treg cells in PBMC will be performed by flow cytometry using appropriate fluorochrome conjugated monoclonal antibodies for CD25 and FoxP3 markers
Identification of T regulatory cells | 3 months post vaccination
  Evaluation of Treg cells in PBMC will be performed by flow cytometry using appropriate fluorochrome conjugated monoclonal antibodies for CD25 and FoxP3 markers
Identification of T regulatory cells | 6 months post vaccination
  Evaluation of Treg cells in PBMC will be performed by flow cytometry using appropriate fluorochrome conjugated monoclonal antibodies for CD25 and FoxP3 markers
Immune response to vaccination | Baseline: at vaccination
  Post-vaccination serum H1N1 antibodies titers (IgG and IgM) will be measured by an ELISA kit
Immune response to vaccination | 3 months post vaccination
  Post-vaccination serum H1N1 antibodies titers (IgG and IgM) will be measured by an ELISA kit
Immune response to vaccination | 6 months post vaccination
  Post-vaccination serum H1N1 antibodies titers (IgG and IgM) will be measured by an ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Francis Corazza, MD, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - HUDERF, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chintagari NR, Nguyen J, Belcher JD, Vercellotti GM, Alayash AI. Haptoglobin attenuates hemoglobin-induced heme oxygenase-1 in renal proximal tubule cells and kidneys of a mouse model of sickle cell disease. Blood Cells Mol Dis. 2015 Mar;54(3):302-6. doi: 10.1016/j.bcmd.2014.12.001. Epub 2014 Dec 22. PMID 25582460
- [Background] Cunnington AJ, Njie M, Correa S, Takem EN, Riley EM, Walther M. Prolonged neutrophil dysfunction after Plasmodium falciparum malaria is related to hemolysis and heme oxygenase-1 induction. J Immunol. 2012 Dec 1;189(11):5336-46. doi: 10.4049/jimmunol.1201028. Epub 2012 Oct 24. PMID 23100518
- [Background] De Montalembert M, Abboud MR, Fiquet A, Inati A, Lebensburger JD, Kaddah N, Mokhtar G, Piga A, Halasa N, Inusa B, Rees DC, Heath PT, Telfer P, Driscoll C, Al Hajjar S, Tozzi A, Jiang Q, Emini EA, Gruber WC, Gurtman A, Scott DA. 13-valent pneumococcal conjugate vaccine (PCV13) is immunogenic and safe in children 6-17 years of age with sickle cell disease previously vaccinated with 23-valent pneumococcal polysaccharide vaccine (PPSV23): Results of a phase 3 study. Pediatr Blood Cancer. 2015 Aug;62(8):1427-36. doi: 10.1002/pbc.25502. Epub 2015 Mar 23. PMID 25810327
- [Background] Hankins J, Jeng M, Harris S, Li CS, Liu T, Wang W. Chronic transfusion therapy for children with sickle cell disease and recurrent acute chest syndrome. J Pediatr Hematol Oncol. 2005 Mar;27(3):158-61. doi: 10.1097/01.mph.0000157789.73706.53. PMID 15750449
- [Background] Lanaro C, Franco-Penteado CF, Albuqueque DM, Saad ST, Conran N, Costa FF. Altered levels of cytokines and inflammatory mediators in plasma and leukocytes of sickle cell anemia patients and effects of hydroxyurea therapy. J Leukoc Biol. 2009 Feb;85(2):235-42. doi: 10.1189/jlb.0708445. Epub 2008 Nov 12. PMID 19004988
- [Background] Lederman HM, Connolly MA, Kalpatthi R, Ware RE, Wang WC, Luchtman-Jones L, Waclawiw M, Goldsmith JC, Swift A, Casella JF; BABY HUG Investigators. Immunologic effects of hydroxyurea in sickle cell anemia. Pediatrics. 2014 Oct;134(4):686-95. doi: 10.1542/peds.2014-0571. Epub 2014 Sep 1. PMID 25180279
- [Background] Mohri T, Ogura H, Koh T, Fujita K, Sumi Y, Yoshiya K, Matsushima A, Hosotsubo H, Kuwagata Y, Tanaka H, Shimazu T, Sugimoto H. Enhanced expression of intracellular heme oxygenase-1 in deactivated monocytes from patients with severe systemic inflammatory response syndrome. J Trauma. 2006 Sep;61(3):616-23; discussion 623. doi: 10.1097/01.ta.0000238228.67894.d7. PMID 16966997
- [Background] Nickel RS, Osunkwo I, Garrett A, Robertson J, Archer DR, Promislow DE, Horan JT, Hendrickson JE, Kean LS. Immune parameter analysis of children with sickle cell disease on hydroxycarbamide or chronic transfusion therapy. Br J Haematol. 2015 May;169(4):574-83. doi: 10.1111/bjh.13326. Epub 2015 Mar 5. PMID 25753210
- [Background] Pathare A, Al Kindi S, Alnaqdy AA, Daar S, Knox-Macaulay H, Dennison D. Cytokine profile of sickle cell disease in Oman. Am J Hematol. 2004 Dec;77(4):323-8. doi: 10.1002/ajh.20196. PMID 15551290
- [Background] Purohit S, Alvarez O, O'Brien R, Andreansky S. Durable immune response to inactivated H1N1 vaccine is less likely in children with sickle cell anemia receiving chronic transfusions. Pediatr Blood Cancer. 2012 Dec 15;59(7):1280-3. doi: 10.1002/pbc.24206. Epub 2012 May 24. PMID 22628221
- [Background] Estcourt LJ, Fortin PM, Hopewell S, Trivella M, Wang WC. Blood transfusion for preventing primary and secondary stroke in people with sickle cell disease. Cochrane Database Syst Rev. 2017 Jan 17;1(1):CD003146. doi: 10.1002/14651858.CD003146.pub3. PMID 28094851
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Yazdanbakhsh K. Mechanisms of sickle cell alloimmunization. Transfus Clin Biol. 2015 Aug;22(3):178-81. doi: 10.1016/j.tracli.2015.05.005. Epub 2015 Jun 6. PMID 26056038